CLINICAL TRIAL: NCT04737798
Title: Comparison of the Effects of Oil Pulling Therapy With Sesame Oil or Coconut Oil Using 4- Day Plaque Regrowth Study Model: A Randomized Crossover Clinical Trial
Brief Title: Comparison of the Effects of Oil Pulling Therapy With Different Oils
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yasemin Sezgin, associate prof, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BaskentU7
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Gingivitis
Keywords: oil pulling; gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Coconut Oil; Sesame Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oil pulling with coconut oil (Experimental): patients used oil pulling therapy with coconut oil for 4 days
  Interventions: Other: oil pulling with coconut oil
- oil pulling with sesame oil (Active Comparator): patients used oil pulling therapy with sesame oil for 4 days
  Interventions: Other: oil pulling with sesame oil

INTERVENTIONS:
Other: oil pulling with coconut oil — using oil pulling therapy with coconut oil
  Arms: oil pulling with coconut oil
Other: oil pulling with sesame oil — using oil pulling therapy with sesame oil
  Arms: oil pulling with sesame oil

SUMMARY:
Oil pulling" or "oil swishing" originates from ancient Ayurvedic medicine in India and now practiced in other parts of the world as a form of complementary and alternative medicine. It has been described as Kavalagraha or Gandhoosha in the ayurvedic texts of Charaka Samhita and Sushruta Samhita. It is a procedure that involves swishing oil in the mouth a period of 15 min, before spitting it out.

In addition to its systemic benefits, oil pulling therapy has also benefits on oral health.

The oil pulling therapy can be performed by using edible oils like sesame oil, sunflower oil and coconut oil. However, there is only one study in the literature comparing the effect of oil pulling therapy using coconut oil versus sesame oil on plaque-induced gingivitis and the results were in favor of coconut oil.

In order to clarify the gap in the literature on this field, this study was designed to compare the plaque-inhibiting effects of oil pulling therapy with sesame oil or coconut oil using 4- day plaque regrowth study model.

DETAILED DESCRIPTION:
The study is conducted as an observer masked, cross over design with a single-center where the participants were randomly allocated to groups. Before the initiation of the study period all participants underwent thorough scaling and polishing of the teeth by both hand and ultrasonic instruments to remove all plaque, calculus and stain and were instructed in how to maintain oral hygiene. This phase considered as a preparatory period by the end of this period all participants obtained healthy gingiva clinically.

The randomization of the participants were provided by closed envelop system (BM). The conductors of the study were blinded to the mouthrinses received by participants. The tested products and regimens of use are shown in Table 1. Identical coded bottles were used to fill the mouthrinses. The bottles also had stickers on explaining the usage instructions. On the first day of each study period, to confirm all patients to have plaque score of 0 at the baseline, erythrosine was applied to all teeth and then scaling and polishing to remove plaque and extrinsic stain and disclosing of the teeth was performed. All tooth cleaning applications (other rinse, chewing gum or toothbrushing / toothpaste) were forbidden for 4 days of study protocol and rinsing regimen was performed. The tested agents included the following: 1) Sesame oil (10 ml, twice daily 15-20 minute) 2) Coconut oil (10 ml, twice daily 15-20 minute). Participants were instructed to perform the mouthrinsing after breakfast and dinner and to avoid rinsing, eating and drinking following hour after rinsing. Even though the mouthrinses were in provided identical bottles and patients were not informed about the products however due to the taste and color differences of the products total subject blindness could not be achieved.

On day 5 (Friday), each subject was scored for staining using Lobene stain index following an oral soft tissue examination. Following the satin scoring erythrosine disclosing was performed and Turesky et al. modification of the Quigley and Hein index was used for plaque scoring. All buccal and lingual surfaces of all fully erupted permanent teeth, with the exception of the third molars were scored for stain and plaque. Six sites of each teeth were also used to score Gingival Index (GI) and bleeding on probing (BOP). All clinical examinations were performed by a single trained and calibrated clinician (YS) who was masked to the study.

Following the recording of clinical parameters, all plaque and tooth stain (if present) were removed by polishing and washout period of 14 days was awaited after the second phase of the study. For the washout period, the subjects were instructed to go on to their routine oral hygiene habits. Following this period the procedures explained before were repeated until each participant used each of the rinses for the second phase of the study.

Standardized questionnaire were filled by the participants in order to evaluate their attitudes and occurrence of adverse effects with regard to the product used at the end of each phase. The questions evaluated the flavor of the mouthrinse, the alteration in the taste of food and drinks, the perception of the plaque reduction, the staining that the mouthrinse created, the feeling to create nausea. Five point Likert type scale was used to collect the responses to the questions which ranged from 1- "very negative" to 5- "very positive" excluding the question about the preference of the product. At the end of each phase participants were asked to bring the bottles to control the remaining mouthrinses in order to control the compliance of the participants.

ELIGIBILITY:
Inclusion Criteria:

* no systemic disease
* having ≥ 22 natural teeth,
* having no removable or fixed prostheses or fixed and removable orthodontic appliances.

Exclusion Criteria:

* use of antibiotics and anti-inflammatory drugs in previous 6 months
* allergy to any ingredient used in the study
* smokers
* pregnant of lactating females
* history of mouthrinses, gels or chewing gums use that contains antimicrobial agents in the preceding 3 months
* having teeth with probing depth ≥4mm and signs of gingival inflammation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
plaque index | day 5
  plaque regrowth inhibition will be tested using the Turesky et al. 21 modification of the Quigley and Hein index.a score of 0 to 5 is assigned to each facial and lingual nonrestored surface of all the teeth except third molars, as follows: 0: No plaque; 1:Separate flecks of plaque at the cervical margin of the tooth; 2:A thin continuos band of plaque (up to one mm) at the cervical margin of the tooth; 3: A band of plaque wider than one mm but covering less than one-third of the crown of the tooth; 4:Plaque covering at least one-third but less than two-thirds of the crown of the tooth; 5: Plaque covering two-thirds or more of the crown of the tooth. An index for the entire mouth is determined by dividing the total score by the number surfaces ( a maximum of 2 x 2 x 14 = 56 surfaces) examined.lower values means that the agent has better plaque inhbiting effect

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Sezgin, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No